CLINICAL TRIAL: NCT01159678
Title: Online Psychoeducation for Sexual Dysfunction in Cancer Survivors
Acronym: OPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Lori Brotto, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H10-01032
Record Dates: First submitted 2010-06-22; First posted 2010-07-09 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- online psychoeducation (Experimental)
  Interventions: Behavioral: online psychoeducation

INTERVENTIONS:
Behavioral: online psychoeducation — The online psychoeducation contains 12 modules which will be administered once per week over the course of three months. The content of each module is as follows:
  1. Important of sexuality to quality of life. & Definitions of sexual desire and arousal.
  2. Consideration of the predisposing, precipitating, and perpetuating factors in his/her sexual difficulties.
  3. Sexual beliefs.
  4. Mindfulness.
  5. Genital anatomy and physiology.
  6. Body Image.
  7. Relationship satisfaction and communication.
  8. Body-oriented mindfulness exercises (focusing and self-observation).
  9. Using Thought records.
  10. Mindfulness and the thought stream.
  11. Sexual aids to boost arousal.
  12. Moving on.
  In addition to these weekly modules, all participants will have access to a moderated and password-protected bulletin board to which participants can post questions and the PI will respond.

SUMMARY:
The purpose of this study is to test an online psychoeducational intervention for men and women with sexual difficulties after surgery for colorectal (men and women) or gynecological (women only) cancer. A psychoeducational intervention is a brief, educational treatment that encourages participants to also pay attention to, and modify, their thoughts, feelings, and behaviour.

DETAILED DESCRIPTION:
Experiencing a diagnosis of cancer may dramatically alter the way a person feels about themselves, their body, and their significant relationships at sexual and intimate levels1. Cancer and its treatments affect the physiological, psychological, and sociological realms of a survivor's life and his/her ability to experience sexual health. Sexual health is recognized as an integral aspect of quality of life (QOL) during cancer and is increasingly receiving research and clinical attention. Sexual changes following the treatment of gynaecologic (i.e.: ovarian, endometrial, cervical) and colorectal cancers are common though often not discussed. Moreover, cancer survivors express dissatisfaction that sexual concerns, and treatment of them, are not discussed in the context of their cancer care. Oncologists frequently are faced with patients inquiring about sexual changes with cancer treatment, but are usually not equipped with accurate and comprehensive data on the precise sexual symptoms to expect or where to refer patients with sexual concerns.

The aims of the study are to assess the efficacy of a 12-module online psychoeducational intervention for sexual health (OPES) on (1) the primary endpoint of sexual distress in male and female cancer survivors with sexual problems; (2) the secondary sexuality-related endpoints of sexual desire, arousal (women) or erection (men), orgasm, and sexual pain; (3) on mood, relationship satisfaction, and quality of life; and (4) to assess gender differences in the proportion of survivors improved on sexual distress.

ELIGIBILITY:
Inclusion Criteria:

1. aged 19-70,
2. treatment of gynaecologic or colorectal cancer by one of the surgical oncologists of the gynaecology or colorectal teams of the BC Cancer Agency centres or satellite sites,
3. received treatment in the past 5 years
4. currently in a relationship
5. currently experiencing sexual dysfunction, and
6. able to participate (both physically and emotionally) in completion of an online psychoeducational treatment.

Exclusion Criteria:

-

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Sexual distress | Questionnaires administered 1 week pre-treatment, 1 week post treatment and six months post treatment
  measured by self report questionnaires

SECONDARY OUTCOMES:
Sexual function | Questionnaires administered 1 week pre-treatment, 1 week post- treatment and six months post treatment
  measured by self-report questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Lori Brotto, PhD, Principal Investigator — University of British Columbia
Locations (1):
- UBC Sexual Health Lab, Vancouver, British Columbia, Canada